CLINICAL TRIAL: NCT03947333
Title: Evaluation of a Patient Portal Intervention for Diabetes: A Two-arm, Parallel-Design, Pilot Randomized Controlled Trial
Brief Title: Evaluation of a Patient Portal Intervention for Diabetes: A Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 190825; 5K23DK106511 (NIH)
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Patient Activation; Patient Web Portals; Health Information Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Patient Participation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients have access to an existing patient web portal (My Health at Vanderbilt) embedded with the My Diabetes Care.
  Interventions: Other: My Diabetes Care
- Control (No Intervention): Patients will have access to an existing patient web portal (My Health at Vanderbilt) NOT embedded with the My Diabetes Care (i.e., usual care).

INTERVENTIONS:
Other: My Diabetes Care — The My Diabetes Care is embedded within an existing patient web portal (My Health at Vanderbilt) and includes graphics to visualize and summarize patients' health data, incorporates motivational strategies (e.g., social comparisons and gamification), provides literacy-level sensitive educational resources, and contains secure-messaging capability.
  Other Names: Patient-facing Diabetes Dashboard
  Arms: Intervention

SUMMARY:
The purpose of this study is to conduct a two-arm, parallel-design, pragmatic randomized controlled trial of a patient portal intervention for diabetes, My Diabetes Care, to evaluate its effect on patient activation and secondary cognitive, behavioral, and clinical outcomes.

DETAILED DESCRIPTION:
300 adult patients with type 2 diabetes mellitus will be randomized to one of two arms. 150 will be assigned to receive access to the intervention (My Diabetes Care) embedded within an existing patient web portal (My Health at Vanderbilt) at Vanderbilt University Medical Center. 150 will be assigned to a usual care comparison arm with access currently available version of My Health at Vanderbilt without the My Diabetes Care. Patients will be invited by mail (or email) to be screened for enrollment in the study. Eligible and interested patients will be emailed a link to a secure study website where they will complete a web consent form. At enrollment, participants will complete a baseline questionnaire and diabetes health data will be abstracted from the patients' electronic health record (EHR) before being randomized to the intervention or control arm. Participants will receive additional follow-up questionnaires and diabetes health data will be abstracted from the EHR at 3-month and 6-month follow-ups to assess outcomes. In addition, system usage will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Currently being treated with at least one antihyperglycemic medication
* Able to speak and read in English
* Reliable access to a computer (desktop or laptop) with internet capabilities
* Active VUMC patient web portal (known as My Health At Vanderbilt) account

Exclusion Criteria:

* Residing in a long term care facility
* Medical condition that affects my memory or ability to think.
* Severe visual impairment
* Currently participating in another diabetes-related research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Martinez W, Hackstadt AJ, Hickson GB, Rosenbloom ST, Elasy TA. Evaluation of the My Diabetes Care Patient Portal Intervention: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 May 25;10(5):e25955. doi: 10.2196/25955. PMID 34032578

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were administratively withdrawn from the study before assignment to groups because they did not complete the baseline study questionnaire (needed prior to randomization). This included 13 patients that could not be reached after enrollment and 4 patients that were reached but did not return the baseline questionnaire. 270 patients completed the baseline study questionnaire and were randomized.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 135 | 135
Completed | 135 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 75 | 152
  >=65 years | 58 | 60 | 118
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 70 | 119
  Male | 83 | 63 | 146
  Other | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 129 | 134 | 263
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 19 | 36
  White | 107 | 111 | 218
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 135 | 135 | 270
Education [Count of Participants; unit: Participants]
  Some high school | 0 | 3 | 3
  High school graduate or GED | 10 | 14 | 24
  Some college or technical school | 41 | 36 | 77
  College graduate (bachelor's degree) | 35 | 35 | 70
  Some graduate work/school | 10 | 11 | 21
  Graduate degree | 38 | 35 | 73
  Unknown or Not Reported | 1 | 1 | 2
Employment [Count of Participants; unit: Participants]
  Working full-time, >=35 hours/week | 54 | 57 | 111
  Working part-time, <35 hours/week | 7 | 7 | 14
  Unemployed or laid off and looking for work | 4 | 4 | 8
  Homemaker | 1 | 1 | 2
  In school | 0 | 1 | 1
  Retired | 57 | 49 | 106
  Disabled, not able to work | 7 | 11 | 18
  Something else | 4 | 4 | 8
  Unknown or Not Reported | 1 | 1 | 2
Insurance [Count of Participants; unit: Participants] — Rows are not mutually exclusive as participants can have more than one type of insurance
  Participants
    Individual Plan: No | 126 | 124 | 250
    Individual Plan: Yes | 9 | 11 | 20
    Group Plan: No | 64 | 67 | 131
    Group Plan: Yes | 71 | 68 | 139
    Governmental Plan: No | 132 | 129 | 261
    Governmental Plan: Yes | 3 | 6 | 9
    Medicaid: No | 134 | 131 | 265
    Medicaid: Yes | 1 | 4 | 5
    Medicare: No | 83 | 78 | 161
    Medicare: Yes | 52 | 57 | 109
    Uninsured: No | 134 | 133 | 267
    Uninsured: Yes | 1 | 2 | 3
Health Literacy [Count of Participants; unit: Participants]
  Adequate | 91 | 87 | 178
  Limited | 43 | 47 | 90
  Unknown or Not Reported | 1 | 1 | 2
Diabetes Duration [Median (Inter-Quartile Range); unit: years] | 12 [7 to 19] | 12 [6 to 19] | 12 [6 to 19]

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Activation at 6 Months
Description: The uni-dimensional, 13-item, Patient Activation Measure (PAM-13) is a valid measure of patient activation (i.e., the knowledge, skills and confidence a person has in managing their own health and health care). Each item uses a 4-point Likert-type scale of response options ranging from strongly disagree to strongly agree. PAM-13 item responses result in total raw scores ranging from 13 to 52, which we converted to the linear interval scale of patient activation scores, ranging from 0 (lowest activation) to 100 (highest activation). The PAM-13 has good psychometric properties including excellent internal consistency reliability (Cronbach's alpha of 0.87). The PAM-13 scores have been used to predict healthcare outcomes including medication adherence and emergency room utilization.
Time Frame: Baseline to 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 135
units on a scale | 4.3 (16.8) | 2.7 (17.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.221, t-test, 1 sided; Mean Difference (Final Values) = 1.6
Statistical Analysis 2: Comparison: Intervention vs Control; Mixed effects model; Test type: Other; p = 0.559, Mixed Models Analysis; fixed-effects estimate of intervention = 0.846, 95% CI 2-sided [-1.99 to 3.68]

2. Primary Outcome: Change in Patient Activation at 3 Months
Description: as for outcome 1
Time Frame: Baseline to 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 135
units on a scale | 3.1 (17.2) | 3.3 (15.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.532, t-test, 1 sided; Mean Difference (Final Values) = -0.2

3. Secondary Outcome: Change in Diabetes Self-Efficacy
Description: The Perceived Diabetes Self-Management Scale (PDSMS) is a valid measure of diabetes self-efficacy (i.e., how confident they feel about their ability to carry out multiple self management tasks). The uni-dimensional, 8-item scale is scored on a five-point Likert scale. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes. PDSMS has excellent internal consistency reliability (Cronbach's alpha of 0.83). PDSMS scores were associated with observed percentage of low blood sugars (r = .21), BMI (r = -.22), percentage of high blood sugars (r = -.36), average blood glucose (r = -.27), and A1C (r = -.25). Thus, the PDSMS appears to be validly associated with important self-management behaviors as well as with indicators of health status and diabetes control.
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the Perceived Diabetes Self-Management Scale (PDSMS) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 134 | 135
units on a scale
  Change at 3 months | 1.0 (4.0) | 0.3 (4.6)
  Change at 6 months | 0.7 (4.9) | 0.8 (5.0)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.086, t-test, 1 sided; Mean Difference (Final Values) = 0.7
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.562, t-test, 1 sided; Mean Difference (Final Values) = -0.1
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.451, Mixed Models Analysis; fixed-effects estimate of intervention = 0.348, 95% CI 2-sided [-0.557 to 1.254]

4. Secondary Outcome: Change in Diabetes Knowledge
Description: The Short Diabetes Knowledge Instrument (SDKI) is a valid measure of diabetes knowledge with an emphasis on controlling blood glucose through diet, recognizing symptoms of abnormal blood glucose, and using healthy eating to prevent complications. It also includes items on foot care and the importance of physical activity for preventing cardiovascular complications. The SDKI is a uni-dimensional, 13-item scale with scores ranging from 0 to 13 (number of items answered correctly). SDKI demonstrated good internal consistency reliability (Cronbach's alpha 0.73) in a multi-ethnic sample of older adults suggesting the instrument can be used to measure diabetes knowledge in diverse populations (Quandt et al. Diabetes Educator, 2014).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the Short Diabetes Knowledge Instrument (SDKI) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 131 | 134
units on a scale
  Change at 3 months | 0.7 (10.3) | -0.1 (10.2)
  Change at 6 months | 2.0 (11.0) | 1.3 (10.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.270, t-test, 1 sided; Mean Difference (Final Values) = 0.8
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.299, t-test, 1 sided; Mean Difference (Final Values) = 0.7
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed effects model; Test type: Other; p = 0.917, Mixed Models Analysis; fixed-effects estimate of intervention = 0.100, 95% CI 2-sided [-1.786 to 1.986]

5. Secondary Outcome: Change in Diabetes Self-Care (General Diet Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA), developed by Toobert and Glasgow (1994), is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The general diet subscale is used to assess general diet adherence. The instrument is based on the self-reported frequency of completing recommended activities during the past 7 days. An example item includes "How often did you follow your recommended diet over the last 7 days?" All responses are converted to percentages. Higher percentages represent better self-care on each subscale. The SDSCA has been used in a number of settings and studies and has been recommended for a standardized evaluation of quality improvement interventions in T2DM in Canada (Majumdar et al., 2005).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the 'general diet' subscale of the Summary of Diabetes Self-Care Activity (SDSCA) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 134
units on a scale
  Change at 3 months | 0.3 (1.6) | 0.1 (1.5)
  Change at 6 months | 0.5 (1.5) | 0.1 (1.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.093, t-test, 1 sided; Mean Difference (Final Values) = 0.2
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.034, t-test, 1 sided; Mean Difference (Final Values) = 0.4
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.103, Mixed Models Analysis; fixed-effects estimate of intervention = 0.242, 95% CI 2-sided [-0.049 to 0.533]

6. Secondary Outcome: Change in Diabetes Self-Care (Specific Diet)
Description: The Summary of Diabetes Self-Care Activity (SDSCA), developed by Toobert and Glasgow (1994), is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The specific diet subscale is used to assess intake of specific foods. The instrument is based on the self-reported frequency of completing recommended activities during the past 7 days. An example item includes "How often did you follow your recommended diet over the last 7 days?" All responses are converted to percentages. Higher percentages represent better self-care on each subscale. The SDSCA has been used in a number of settings and studies and has been recommended for a standardized evaluation of quality improvement interventions in T2DM in Canada (Majumdar et al., 2005).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the 'specific diet' subscale of the Summary of Diabetes Self-Care Activity (SDSCA) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 134
units on a scale
  Change at 3 months | 0.2 (1.6) | 0 (1.3)
  Change at 6 months | 0.3 (1.3) | -0.1 (1.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.116, t-test, 1 sided; Mean Difference (Final Values) = 0.2
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority; p = 0.009, t-test, 1 sided; Mean Difference (Final Values) = 0.4
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.178, Mixed Models Analysis; fixed-effects estimate of intervention = 0.183, 95% CI 2-sided [-0.084 to 0.451]

7. Secondary Outcome: Change in Diabetes Self-Care (Exercise Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA), developed by Toobert and Glasgow (1994), is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The exercise subscale is used to assess exercise adherence. The instrument is based on the self-reported frequency of completing recommended activities during the past 7 days. An example item includes "How often did you follow your recommended diet over the last 7 days?" All responses are converted to percentages. Higher percentages represent better self-care on each subscale. The SDSCA has been used in a number of settings and studies and has been recommended for a standardized evaluation of quality improvement interventions in T2DM in Canada (Majumdar et al., 2005).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the 'exercise' subscale of the Summary of Diabetes Self-Care Activity (SDSCA) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 132
units on a scale
  Change at 3 months | 0.2 (1.6) | -0.1 (1.6)
  Change at 6 months | 0 (1.6) | 0.1 (1.7)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.188, t-test, 1 sided; Mean Difference (Final Values) = 0.2
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.749, t-test, 1 sided; Mean Difference (Final Values) = -0.1
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.847, Mixed Models Analysis; fixed-effects estimate of intervention = 0.031, 95% CI 2-sided [-0.288 to 0.351]

8. Secondary Outcome: Change in Diabetes Self-Care (Self-Monitoring of Blood Glucose Adherence)
Description: The Summary of Diabetes Self-Care Activity (SDSCA), developed by Toobert and Glasgow (1994), is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The blood-glucose testing subscale is used to assess self-monitoring of blood glucose adherence. The instrument is based on the self-reported frequency of completing recommended activities during the past 7 days. An example item includes "How often did you follow your recommended diet over the last 7 days?" All responses are converted to percentages. Higher percentages represent better self-care on each subscale. The SDSCA has been used in a number of settings and studies and has been recommended for a standardized evaluation of quality improvement interventions in T2DM in Canada (Majumdar et al., 2005).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: The blood-glucose testing subscale was administered only to patients that reported testing their blood sugar at home. Participants with missing responses to items on the 'blood-glucose testing' subscale of the Summary of Diabetes Self-Care Activity (SDSCA) were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 118 | 114
units on a scale
  Change at 3 months | 0.3 (2.0) | 0.1 (1.7)
  Change at 6 months | 0.3 (2.1) | 0.1 (1.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.182, t-test, 1 sided; Mean Difference (Final Values) = 0.2
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.158, t-test, 1 sided; Mean Difference (Final Values) = 0.3
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.612, Mixed Models Analysis; fixed-effects estimate of intervention = 0.107, 95% CI 2-sided [-0.305 to 0.519]

9. Secondary Outcome: Change in Diabetes Self-Care (Diabetes Medication Adherence)
Description: The Adherence to Refills and Medications Scale-Diabetes (ARMS-D) is a reliable and valid measure of diabetes medication adherence. The 11-item ARMS-D has good internal consistency reliability (α=0.86). Responses range from 1="none of the time" to 4="all of the time," and are summed to produce an overall adherence score ranging from 12-48, with higher scores representing more problems with medication adherence.
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the Adherence to Refills and Medications Scale-Diabetes (ARMS-D) scale were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 132 | 133
units on a scale
  Change at 3 months | -0.3 (2.0) | 0.2 (1.8)
  Change at 6 months | -0.3 (2.9) | -0.1 (1.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.970, t-test, 1 sided; Mean Difference (Final Values) = -0.5
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.786, t-test, 1 sided; Mean Difference (Final Values) = -0.2
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.670, Mixed Models Analysis; fixed-effects estimate of intervention = -0.088, 95% CI 2-sided [-0.493 to 0.317]

10. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. The five-item, uni-dimensional scale has scores that range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress. The PAID-5 has excellent excellent internal consistency reliability (Cronbach's alpha 0.86) and is associated with measures of depression and hemoglobin A1c.
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the Problem Areas in Diabetes Scale (PAID-5) scale were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 134 | 133
units on a scale
  Change at 3 months | -0.2 (2.8) | -0.2 (3.4)
  Change at 6 months | -0.4 (3.4) | -0.2 (2.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Change at 3 months; Test type: Superiority; p = 0.478, t-test, 1 sided; Median Difference (Final Values) = 0.0
Statistical Analysis 2: Comparison: Intervention vs Control; Change at 6 months; Test type: Superiority; p = 0.666, t-test, 1 sided; Mean Difference (Net) = -0.2
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed Effects Model; Test type: Other; p = 0.601, Mixed Models Analysis; fixed-effects estimate of intervention = -0.150, 95% CI 2-sided [-0.713 to 0.413]

11. Secondary Outcome: Change in Blood Glucose Control
Description: Participants' most recent hemoglobin A1C will be abstracted from participants' electronic medical record at enrollment (T0) and 6 month follow-up (T3).
Time Frame: Baseline to 6-month follow-up
Population: If date of the most recent hemoglobin A1c abstracted from the participant's electronic health record at 6 month follow-up was less than 90 or greater than 365 days from the date of the most recent hemoglobin A1c abstracted from the participant's electronic health record at baseline, then the participant was not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 132
percentage of glycated hemoglobin | 0.1 (1.2) | 0.1 (0.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.654, t-test, 1 sided; Mean Difference (Final Values) = 0.06

12. Secondary Outcome: Change in Blood Pressure Control
Description: Participants' most recent blood pressure measurement will be abstracted from participants' electronic medical record at enrollment (T0) and 6 month follow-up (T3) and will be used to calculate the participants' mean arterial pressure (MAP) using the following formula: MAP = diastolic pressure + 1/3(systolic pressure - diastolic pressure).
Time Frame: Baseline to 6-month follow-up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 135
mmHg | -0.2 (6.9) | -0.2 (7.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.485, t-test, 1 sided; Mean Difference (Final Values) = -0.04

13. Secondary Outcome: Change in Flu Vaccination Status for 2019-20 Flu Season
Description: The participants' influenza vaccination status (vaccinated vs unvaccinated) for the 2019-20 Flu Season will be abstracted from participants' electronic medical record at enrollment (T0), 3 month follow-up (T1).
Time Frame: Baseline, 3-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 135
Participants
  Baseline: Unvaccinated | 42 | 38
  Baseline: Vaccinated | 93 | 97
  3 month follow-up: Unvaccinated | 40 | 33
  3 month follow-up: Vaccinated | 95 | 102
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.480, McNemar
Statistical Analysis 2: Comparison: Control; Test type: Other; p = 0.023, McNemar

14. Secondary Outcome: Change in Low Density Lipoprotein
Description: Participants' most recent low density lipoprotein measurement will be abstracted from participants' electronic medical record at enrollment (T0) and 6 month follow-up (T3).
Time Frame: Baseline to 6-month follow-up
Population: If date of the most recent low density lipoprotein (LDL) abstracted from the participant's electronic health record at 6 month follow-up was less than 90 or greater than 365 days from the date of the most recent LDL abstracted from the participant's electronic health record at baseline, then the participant was not included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 131 | 125
mg/dL | -3.0 (22.7) | -3.8 (36.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.542, t-test, 1 sided; Mean Difference (Final Values) = 0.8

15. Secondary Outcome: Satisfaction/Usability of My Health at Vanderbilt (for Control Group)
Description: The System Usability Scale (SUS) is a valid measure of usability and assesses users' perceptions of ease of use, likability of the interface, and overall satisfaction using a 5- point Likert scale (strongly disagree to strongly agree). The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 85 or above suggests excellent usability. The SUS has been used in several studies of patient facing health information technology (the article describing its psychometric properties has been cited over 500 times) and has excellent internal consistency reliability (Cronbach's alpha of 0.91).
Time Frame: Baseline, 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the System Usability Scale (SUS) were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control
Number analyzed (Participants) | 131
score on a scale
  Baseline | 79.0 (12.9)
  3 month follow-up | 82.4 (13.4)
  6 month follow-up | 83.2 (12.7)

16. Secondary Outcome: Satisfaction/Usability of My Diabetes Care (for Intervention Group)
Description: as for outcome 15
Time Frame: 3-month follow up, 6-month follow-up
Population: Participants with missing responses to items on the System Usability Scale (SUS) were not analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 134
score on a scale
  3 month follow-up | 73.7 (14.3)
  6 month follow-up | 71.7 (15.1)

17. Secondary Outcome: System Usage Data for My Diabetes Care - Total Sessions (Intervention Group Only)
Description: Self-reported system usage will include: participants' total number of visits, total duration of visits, and utilization of embedded features and functionality
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 135
Participants
  None | 12
  One to three | 60
  Four to six | 39
  Seven to nine | 9
  Ten or more | 9
  Unknown or Not Reported | 6

18. Secondary Outcome: System Usage Data for My Diabetes Care - Total Duration of Visits (Intervention Group Only)
Description: as for outcome 17
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 135
Participants
  5 minutes or less | 22
  6 to 10 minutes | 37
  11 to 15 minutes | 21
  16 to 20 minutes | 22
  More than 20 minutes | 15
  Unknown or Not Reported | 18

19. Secondary Outcome: System Usage Data for My Diabetes Care - Utilization of Embedded Features and Functionality (Intervention Group Only)
Description: as for outcome 17
Time Frame: 6-month follow-up
Population: My Diabetes Care features used at least once by the participant. Rows are not mutually exclusive as participants can use more than one feature. Participants with no response to this questionnaire item were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 129
Participants
  Links to information about diabetes: No | 67
  Links to information about diabetes: Yes | 62
  Message your Doctor button: No | 98
  Message your Doctor button: Yes | 31
  Online Patient Support Community button: No | 119
  Online Patient Support Community button: Yes | 10
  Hover over text or icon for more information about your diabetes health data: No | 70
  Hover over text or icon for more information about your diabetes health data: Yes | 59
  Diabetes News Feeds (Diabetes Views or ADA Diabetes Blog): No | 104
  Diabetes News Feeds (Diabetes Views or ADA Diabetes Blog): Yes | 25
  None of the above: No | 99
  None of the above: Yes | 30

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135
Other Adverse Events (participants affected / at risk) | 0/135 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03947333/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03947333/ICF_002.pdf